CLINICAL TRIAL: NCT01331538
Title: Correlation Between Temporomandibular Dysfunction and Cervical Posture in Different Occlusal Angle Classes in Adolescents
Brief Title: Temporomandibular Dysfunction and Cervical Posture
Status: Completed | Type: Observational
Sponsor: University of Nove de Julho (Other)
Responsible Party: Lara Jansiski Motta, Nove de Julho University
Other Study IDs: 82622/08
Record Dates: First submitted 2011-04-06; First posted 2011-04-08 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2009-02

CONDITIONS: Temporomandibular Dysfunction
Keywords: temporomandibular dysfunction; posture
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- adolescents with TMD: adolescents with temporomandibular dysfunction
- No TMD: adolescents without temporomandibular dysfunction

SUMMARY:
The aim of this research was to determine the existence of a correlation between the degree of temporomandibular dysfunction and cervical posture in different occlusal classes in adolescents. A cross-section, observational study was carried out, in which 296 adolescents took part. For the evaluation, the patients were divided into groups according to the presence and severity of the temporomandibular dysfunction, using a questionnaire and occlusal Angle classification. The posture analysis was carried out using photogrammetry and the software Alcimage® to measure the predefined angle based on the protuberances of the Spinous Process of the 7th Cervical Vertebra (C7), Manubrium of the sternum and Mentum Vertex.

DETAILED DESCRIPTION:
The evaluation of signs and symptoms of TMD was obtained from a Questionnaire (15) which includes information regarding difficulties opening the mouth and movement of the mandible, pains in the head, nape of the neck, neck or joint regions, noise in the temporomandibular joints, and the habit of clenching or grinding the teeth. The questionnaire is comprised of 10 questions with possible answers of yes (10 points), sometimes (5 points) and no (0 points). For each question, only one answer can be checked. The total score is used to classify the severity of the TMD as severe (70 to 100 points), moderate (45 to 65), mild (20 to 40) and no dysfunction (0 to 15).

The clinical (visual) assessment of head posture was conducted using a postural grid. Each subject was asked to remain in his or her normal posture, in a standing position. The self balance position was used to standardize the posture of each subject, asking them to look straight ahead, parallel to the floor, keeping the gaze horizontal

ELIGIBILITY:
Inclusion Criteria:

* adolescents, aged between 10 and 20 years. As criteria for inclusion, age group and the presence of first permanent molar

Exclusion Criteria:

* Individuals undergoing orthodontic treatment, those with absent first molars and cases where it was impossible to clinically evaluate the occlusion were excluded.

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: adolescents aged between 10 and 20 years. As criteria for inclusion, age group and the presence of first permanent molar
Sampling Method: Non-Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2009-02; Primary Completion 2009-10 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lara Motta, Ms, Principal Investigator — Nove de Julho University
Locations (1):
- Nove de Julho University, São Paulo, São Paulo, Brazil